CLINICAL TRIAL: NCT01075191
Title: PMOS: Kaletra Double Protease Inhibitors
Brief Title: Kaletra: Therapy With Double Protease Inhibitors
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P05-103
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: Viral load; Resistance; Double protease inhibitors; Mutations; Immune system; Infection; Nucleoside Reverse Transcriptase Inhibitors-free; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected participants: HIV-infected participants taking lopinavir/ritonavir (Kaletra) and one other protease inhibitor.
  Lopinavir/ritonavir (Kaletra) dosing and administration according to the Summary of Product Characteristics (three 133 mg/33 mg capsules twice daily or two 200 mg/50 mg tablets twice daily).

SUMMARY:
Therapy with lopinavir/ritonavir (Kaletra) and one other protease inhibitor in Human Immunodeficiency Virus participants

DETAILED DESCRIPTION:
This study is intended to observe and collect data on the usage, dosing, tolerability, and effectiveness of lopinavir/ritonavir (Kaletra) when used as part of a Nucleoside Reverse Transcriptase Inhibitors-free double protease regimen. Enrollment in the study was independent of the decision to prescribe Kaletra.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Human Immunodeficiency Virus infection
* Participants on lopinavir/ritonavir (Kaletra) and one other protease inhibitor

Exclusion Criteria:

* Hypersensitivity against lopinavir, ritonavir or other ingredients
* Severe liver insufficiency
* No concomitant astemizole, terfenadine, oral midazolam, triazolam, cisapride, pimozide, amiodarone, ergotamine, dihydroergotamine, ergometrine, methylergometrine, vardenafil and St. John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample; Human Immunodeficiency Virus-infected participants
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2004-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Simianer, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department
Locations (17):
- Germany (17):
  - Site Reference ID/Investigator# 48283, Berlin
  - Site Reference ID/Investigator# 28131, Berlin
  - Site Reference ID/Investigator# 66422, Berlin
  - Site Reference ID/Investigator# 28123, Berlin
  - Site Reference ID/Investigator# 28109, Berlin
  - Site Reference ID/Investigator# 28115, Dortmund
  - Site Reference ID/Investigator# 28124, Frankfurt
  - Site Reference ID/Investigator# 28127, Frankfurt
  - Site Reference ID/Investigator# 28119, Frankfurt
  - Site Reference ID/Investigator# 5318, Krefeld
  - Site Reference ID/Investigator# 28112, Ludwigshafen
  - Site Reference ID/Investigator# 28118, Munich
  - Site Reference ID/Investigator# 28113, Munich
  - Site Reference ID/Investigator# 28111, Münster
  - Site Reference ID/Investigator# 28129, Münster
  - Site Reference ID/Investigator# 28133, Stuttgart
  - Site Reference ID/Investigator# 28126, Wuppertal

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-infected Participants: HIV-infected participants taking lopinavir/ritonavir (Kaletra) and one other protease inhibitor.
  Lopinavir/ritonavir (Kaletra) dosing and administration according to the Summary of Product Characteristics (3 capsules twice daily or 2 tablets twice daily).
Period: Overall Study
Arm/Group | HIV-infected Participants
Started | 60 (65 participants were enrolled; 5 protocol violations were excluded from all analyses except safety.)
Discontinued Year 1 | 7
Discontinued Year 2 | 6
Discontinued Year 3 | 5
Completed | 42
Not Completed | 18
Not completed — Death | 1
Not completed — Intensification | 3
Not completed — Co-morbidities | 1
Not completed — Adverse Event | 4
Not completed — Noncompliance | 3
Not completed — Therapy Break | 3
Not completed — Patient's Wish | 2
Not completed — Unknown Reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: years] — In 10 participants, age was missing.
  years | 44.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 53
Region of Enrollment [Number; unit: participants]
  Germany | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus -1 Ribonucleic Acid (HIV-1 RNA) <50 Copies/mL
Description: Viral load (number of HIV-1 RNA copies in the blood) was measured at baseline and scheduled study visits. A decrease in viral load is a measure used to assess the effectiveness of antiviral treatments. The percentage of participants with HIV RNA less than 50 copies/mL at each time point is presented.
Time Frame: Baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
Population: Evaluable participants. n=number of evaluable participants with given measurement at time point.
Measure: Number; unit: percentage of participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 60
percentage of participants
  Baseline (n=58) | 8.6
  Week 4 (n=42) | 26.2
  Week 12 (n=50) | 40.0
  Week 24 (n=48) | 56.3
  Week 36 (n=42) | 69.1
  Week 48 (n=41) | 65.9
  Week 60 (n=38) | 68.4
  Week 72 (n=38) | 76.3
  Week 84 (n=34) | 76.5
  Week 96 (n=30) | 56.7
  Week 108 (n=34) | 58.8
  Week 120 (n=30) | 63.3
  Week 132 (n=31) | 58.1
  Week 144 (n=29) | 69.0

2. Secondary Outcome: Change From Baseline in Absolute CD4 Cell Count
Description: Increases in CD4 count are a biomarker for antiretroviral treatment effectiveness in restoring immunologic function. Changes in participants' CD4-positive (CD4+) T-lymphocyte counts were assessed by measuring the change from Baseline in the number of CD4+ cells at scheduled study visits.
Time Frame: Baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
Population: Evaluable participants. n=number of evaluable participants with given measurement at time point.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 60
cells/µL
  Baseline (n=58) | 312.0 (227)
  Change at Week 4 (n=44) | 48.2 (134)
  Change at Week 12 (n=51) | 115.7 (186)
  Change at Week 24 (n=48) | 124.5 (176)
  Change at Week 36 (n=43) | 122.6 (216)
  Change at Week 48 (n=42) | 129.0 (247)
  Change at Week 60 (n=38) | 155.4 (267)
  Change at Week 72 (n=38) | 180.8 (200)
  Change at Week 84 (n=33) | 225.7 (217)
  Change at Week 96 (n=30) | 227.7 (210)
  Change at Week 108 (n=35) | 274.7 (244)
  Change at Week 120 (n=30) | 274.3 (284)
  Change at Week 132 (n=31) | 260.8 (214)
  Change at Week 144 (n=28) | 271.8 (232)

3. Secondary Outcome: Change From Baseline in Relative CD4 Cell Count
Description: Increases in relative CD4 count (the percentage of total lymphocytes that are CD4 cells) are a biomarker for antiretroviral treatment effectiveness in restoring immunologic function. Changes in participants' CD4-positive (CD4+) T-lymphocyte counts were assessed by measuring the change from Baseline in the percentage of CD4+ cells at scheduled study visits.
Time Frame: Baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
Population: Evaluable participants. n=number of evaluable participants with given measurement at time point.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 60
percentage of cells
  Baseline (n=59) | 16.8 (9.4)
  Change at Week 4 (n=42) | 1.4 (3.3)
  Change at Week 12 (n=45) | 2.8 (5.2)
  Change at Week 24 (n=42) | 4.1 (5.6)
  Change at Week 36 (n=38) | 4.9 (7.0)
  Change at Week 48 (n=35) | 4.9 (6.7)
  Change at Week 60 (n=32) | 5.4 (6.2)
  Change at Week 72 (n=32) | 5.0 (6.4)
  Change at Week 84 (n=28) | 5.7 (6.4)
  Change at Week 96 (n=24) | 6.3 (5.3)
  Change at Week 108 (n=28) | 7.9 (7.4)
  Change at Week 120 (n=24) | 7.6 (9.0)
  Change at Week 132 (n=25) | 8.4 (8.9)
  Change at Week 144 (n=23) | 8.6 (8.0)

4. Secondary Outcome: Change From Baseline in Absolute CD8 Cell Count
Description: Decreases in CD8 count are a biomarker for antiretroviral treatment effectiveness in restoring immunologic function. Changes in participants' CD8-positive (CD8+) T-lymphocyte counts were assessed by measuring the change from Baseline in the number of CD8+ cells at scheduled study visits.
Time Frame: Baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
Population: Evaluable participants. n=number of evaluable participants with given measurement at time point.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 60
cells/µL
  Baseline (n=60) | 1180.8 (713)
  Change at Week 4 (n=44) | 109 (728)
  Change at Week 12 (n=51) | 195 (762)
  Change at Week 24 (n=49) | 66 (671)
  Change at Week 36 (n=43) | -59 (774)
  Change at Week 48 (n=42) | -105 (777)
  Change at Week 60 (n=38) | -42 (706)
  Change at Week 72 (n=38) | 4 (676)
  Change at Week 84 (n=33) | 132 (637)
  Change at Week 96 (n=30) | 54 (616)
  Change at Week 108 (n=35) | 39 (529)
  Change at Week 120 (n=30) | 24 (721)
  Change at Week 132 (n=31) | -57 (676)
  Change at Week 144 (n=28) | -3 (644)

5. Secondary Outcome: Change From Baseline in Relative CD8 Cell Count
Description: Decreases in relative CD8 count (the percentage of total lymphocytes that are CD8 cells) are a biomarker for antiretroviral treatment effectiveness in restoring immunologic function. Changes in participants' CD8-positive (CD8+) T-lymphocyte counts were assessed by measuring the change from Baseline in the percentage of CD8+ cells at scheduled study visits.
Time Frame: Baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
Population: Evaluable participants. n=number of evaluable participants with given measurement at time point.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 60
percentage of cells
  Baseline (n=59) | 60.4 (15.0)
  Change at Week 4 (n=41) | -2.2 (13.9)
  Change at Week 12 (n=45) | -2.1 (15.8)
  Change at Week 24 (n=42) | -7.1 (11.6)
  Change at Week 36 (n=38) | -8.2 (12.1)
  Change at Week 48 (n=35) | -8.6 (12.1)
  Change at Week 60 (n=32) | -11.0 (9.4)
  Change at Week 72 (n=31) | -10.9 (12.4)
  Change at Week 84 (n=28) | -10.7 (13.3)
  Change at Week 96 (n=24) | -10.0 (12.7)
  Change at Week 108 (n=28) | -13.2 (13.0)
  Change at Week 120 (n=24) | -11.5 (13.4)
  Change at Week 132 (n=25) | -13.1 (12.8)
  Change at Week 144 (n=23) | -13.5 (13.4)

6. Secondary Outcome: Change From Baseline in CD4/CD8 T-cell Ratio
Description: The CD4/CD8 T-cell ratio, also known as the T-lymphocyte helper/suppressor profile, presents the number of lymphocytes in the blood positive for CD4 cells compared with the number positive for CD8 cells. Changes in participants' CD4/CD8 T-lymphocyte ratio were assessed by measuring the change from Baseline in the ratio at scheduled study visits.
Time Frame: Baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
Population: Evaluable participants. n=number of evaluable participants with given measurement at time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 60
ratio
  Baseline (n=60) | 0.3 (0.2)
  Change at Week 4 (n=44) | 0.1 (0.1)
  Change at Week 12 (n=51) | 0.1 (0.2)
  Change at Week 24 (n=48) | 0.1 (0.2)
  Change at Week 36 (n=43) | 0.2 (0.3)
  Change at Week 48 (n=42) | 0.2 (0.3)
  Change at Week 60 (n=38) | 0.3 (0.3)
  Change at Week 72 (n=38) | 0.2 (0.3)
  Change at Week 84 (n=33) | 0.3 (0.3)
  Change at Week 96 (n=30) | 0.2 (0.2)
  Change at Week 108 (n=35) | 0.3 (0.3)
  Change at Week 120 (n=30) | 0.3 (0.3)
  Change at Week 132 (n=31) | 0.3 (0.3)
  Change at Week 144 (n=28) | 0.3 (0.4)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Serious Adverse Events (SAEs) and Adverse Events (AEs) were reported by the investigators using standard reporting forms and were sent directly to the sponsor's pharmacovigilance department.
Groups:
- HIV-infected Participants: HIV-infected patients taking lopinavir/ritonavir (Kaletra) and one other protease inhibitor.
  Lopinavir/ritonavir (Kaletra) dosing and administration according to the Summary of Product Characteristics (3 capsules twice daily or 2 tablets twice daily).
  Safety data presents all enrolled participants, including 5 protocol violations.
Arm/Group | HIV-infected Participants
Serious Adverse Events (participants affected / at risk) | 4/65
Other Adverse Events (participants affected / at risk) | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-infected Participants (N=65)
Urosepsis (Renal and urinary disorders) | 1
Gastroenteritis clostridial (Gastrointestinal disorders) | 1
Hepatitis C (Infections and infestations) | 1
Anal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — leading to death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.